CLINICAL TRIAL: NCT05658939
Title: Safety and Effectiveness of Integrative Korean Medicine Treatment for Traffic Accident During Pregnancy : Retrospective Chart Review Study and Survey Research
Brief Title: Safety and Effectiveness of Integrative Korean Medicine Treatment for Traffic Accident During Pregnancy
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2022-05
Record Dates: First submitted 2022-11-09; First posted 2022-12-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Traffic Accident

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Phone/Internet survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone/internet for patients.

SUMMARY:
The purpose of this study is to reveal the efficacy and safety of integrative korean medicine treatment for pregnant women who suffered a traffic accident. A retrospective chart review and follow-up were conducted.

From January 1, 2018 to April 22, 2022, pregnant women who visited an korean medicine hospital due to a traffic accident were subjected to a retrospective study of patient medical records and follow-up.

DETAILED DESCRIPTION:
Medical records of selected patients will be analyzed, and telephone or internet surveys will be conducted for each patient. The survey questions are Numeric rating scale(NRS), Neck disability index(NDI) score, Oswestry Disability Index(ODI) score, Shoulder Pain and Disability Index(SPADI) score, The Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) score, EuroQol 5-dimension 5-level(EQ-5D-5L) score and patient global impression of change (PGIC) score, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visited hospital due to symptoms caused by a traffic accident during pregnancy and received one or more korean medicine treatment as an inpatient or outpatient treatment
* Patients who understand the purpose and contents of the study and agree to participate in the study
* Patients with communication skills and mental/physical ability to respond appropriately to questionnaires

Exclusion Criteria:

* Patients under the age of 18 at the time of the first visit
* Patients who received treatment without being aware of pregnancy
* Patients who have undergone only consultation or Western treatment at the hospital
* Patients whose participation in the study is difficult for the researcher to judge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 1, 2018 to April 22, 2022, patients who visited Daejeon Jasaeng Korean Medicine Hospital due to a traffic accident during pregnancy were included.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Effectiveness Outcome : Numeric rating scale (NRS) | Finish survey by August 2022
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS scores were collected for each patient's chief complaints. For outpatients, the NRS scores on the first and last outpatient visit days, and for inpatients, the NRS scores on the day of admission and discharge were collected through the electronic medical records(EMRs). In the follow-up questionnaire, the current NRS score was also collected for each patient's chief complaints.

SECONDARY OUTCOMES:
Effectiveness Outcome : Neck Disability Index (NDI) | Finish survey by August 2022
  The NDI questionnaire is a 10-item questionnaire designed to evaluate functional disorders related to the cervical spine. Each item consists of 6 levels ranging from 0 to 5, and the higher the score, the more severe the functional impairment.
Effectiveness Outcome : Oswestry Disability Index (ODI) | Finish survey by August 2022
  The ODI is a 10-item questionnaire developed to evaluate the degree of disability for low back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean ODI questionnaire.
Effectiveness Outcome : Shoulder Pain and Disability Index (SPADI) | Finish survey by August 2022
  The SPADI is a questionnaire designed to evaluate functional impairments related to the shoulder and consists of two dimensions: the pain dimension, 5 questions; the functional activities, 8 questions. Each item consists of 0-10 points, and the higher the score, the more severe the shoulder dysfunction.
Effectiveness Outcome : The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Finish survey by August 2022
  The WOMAC is a questionnaire evaluation tool designed to evaluate the joint function of the knee joint and consists of three subscales: pain, 5 questions; stiffness, 2 questions; physical function, 17 questions. Each item consists of 1-5 points, and the higher the score, the worse the condition of the knee joint.
Effectiveness Outcome : EuroQol 5-dimension 5-level (EQ-5D-5L) | Finish survey by August 2022
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used
Effectiveness Outcome : Patient Global Impression of Change (PGIC) | Finish survey by August 2022
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).

OTHER OUTCOMES:
Survey ( Obstetric and neonatal outcomes checklist) | Finish survey by August 2022
  Obstetric and neonatal outcomes
Number of participants with Symptoms related/not related to pregnancy | Finish survey by August 2022
  Symptoms related/not related to pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Sunah Kim, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No